CLINICAL TRIAL: NCT00812175
Title: Global Investigation of Therapeutic Decisions in Hepatocellular Carcinoma and of Its Treatment With Sorafenib
Acronym: GIDEON
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13414; NX0802 (Other: company internal)
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; HCC; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Systemic oral therapy according to product information

SUMMARY:
In this international non-interventional study safety and clinical data concerning the treatment of patients suffering from Hepatocellular Carcinoma (HCC) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with histologically/cytologically documented or radiographically diagnosed unresectable HCC who are candidates for systemic therapy and for whom a decision to treat with Nexavar has been made. Radiographic diagnosis HCC NIS, needs typical findings of HCC by radiographic method i.e. on multi-dimensional, dynamic CT, CT hepatic arteriography (CTHA)/CT arterial portography (CTAP), or MRI.
* Patients must have signed an informed consent form
* Patients must have a life expectancy of at least 8 weeks

Exclusion Criteria:

* Exclusion criteria must follow the approved local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable HCC who are candidates for systemic therapy and in whom a decision to treat with Nexavar has been made under real-life practice conditions and in a variety of patient subsets.
Sampling Method: Non-Probability Sample
Enrollment: 3371 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The safety of Nexavar in all patients with unresectable HCC who are candidates for systemic therapy and in whom a decision to treat with Nexavar has been made under real-life practice conditions | at each follow-up visit, every 2-4 months on average

SECONDARY OUTCOMES:
Efficacy [overall survival (OS), progression-free survival (PFS), time to progression (TTP), response rate (RR), stable disease(SD) rate] by the Response Evaluation Criteria in Solid Tumor (RECIST) Criteria of Nexavar | at every visit, roughly every 2-4 months
The duration of therapy with Nexavar in a variety of settings according to patient characteristics and other variables | at every visit, roughly every 2-4 months
To evaluate the methods of patient evaluation, diagnosis and follow up | at every visit, roughly every 2-4 months
To evaluate the co-morbidities in patients with unresectable HCC and their influence on treatment and outcome | at every visit, roughly every 2-4 months
To evaluate the practice patterns of the physicians involved in the care of patients with HCC under real-life conditions | at every visit, roughly every 2-4 months
Reports of adverse events | at every visit, roughly every 2-4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (75):
- United States (37):
  - Many Locations, Alabama
  - Many Locations, Arizona
  - Many Locations, Arkansas
  - Many Locations, California
  - Many Locations, Colorado
  - Many Locations, Connecticut
  - Many Locations, Florida
  - Many Locations, Georgia
  - Many Locations, Hawaii
  - Many Locations, Illinois
  - Many Locations, Indiana
  - Many Locations, Iowa
  - Many Locations, Kansas
  - Many Locations, Kentucky
  - Many Locations, Louisiana
  - Many Locations, Maryland
  - Many Locations, Massachusetts
  - Many Locations, Michigan
  - Many Locations, Minnesota
  - Many Locations, Missouri
  - Many Locations, Nebraska
  - Many Locations, Nevada
  - Many Locations, New Hampshire
  - Many Locations, New Jersey
  - Many Locations, New York
  - Many Locations, North Carolina
  - Many Locations, Ohio
  - Many Locations, Oklahoma
  - Many Locations, Oregon
  - Many Locations, Pennsylvania
  - Many Locations, South Carolina
  - Many Locations, Tennessee
  - Many Locations, Texas
  - Many Locations, Utah
  - Many Locations, Virginia
  - Many Locations, Washington
  - Many Locations, Wisconsin
- Many Locations, Canada
- Many Locations, China
- Many Locations, Colombia
- Many Locations, Croatia
- Many Locations, Czechia
- Many Locations, Finland
- Many Locations, France
- Many Locations, Greece
- Many Locations, Hong Kong
- Many Locations, Hungary
- Many Locations, India
- Many Locations, Indonesia
- Many Locations, Israel
- Many Locations, Italy
- Many Locations, Japan
- Many Locations, Kazakhstan
- Many Locations, Libya
- Many Locations, Malaysia
- Many Locations, Mexico
- Many Locations, Norway
- Many Locations, Pakistan
- Many Locations, Philippines
- Many Locations, Portugal
- Many Locations, Qatar
- Many Locations, Romania
- Many Locations, Russia
- Many Locations, Singapore
- Many Locations, Slovakia
- Many Locations, South Korea
- Many Locations, Spain
- Many Locations, Sweden
- Many Locations, Syria
- Many Locations, Thailand
- Many Locations, Ukraine
- Many Locations, United Arab Emirates
- Many Locations, Uruguay
- Many Locations, Venezuela
- Many Locations, Vietnam

REFERENCES:
- [Result] Ye SL, Chen X, Yang J, Bie P, Zhang S, Liu F, Liu L, Zhou J, Dou K, Hao C, Shao G, Xia Q, Chen Y, Yang J, Deng X, Liu Y, Yuan Y, Fu Z, Nakajima K, Yip CS, Lu Z. Safety and efficacy of sorafenib therapy in patients with hepatocellular carcinoma: final outcome from the Chinese patient subset of the GIDEON study. Oncotarget. 2016 Feb 9;7(6):6639-48. doi: 10.18632/oncotarget.6781. PMID 26735891
- [Derived] Ye SL, Yang J, Bie P, Zhang S, Chen X, Liu F, Liu L, Zhou J, Dou K, Hao C, Shao G, Xia Q, Chen Y, Yang J, Deng X, Liu Y, Yuan Y, Fu Z, Nakajima K, Lv Z. Safety assessment of sorafenib in Chinese patients with unresectable hepatocellular carcinoma: subgroup analysis of the GIDEON study. BMC Cancer. 2018 Mar 2;18(1):247. doi: 10.1186/s12885-018-4144-9. PMID 29499662
- [Derived] Kudo M, Lencioni R, Marrero JA, Venook AP, Bronowicki JP, Chen XP, Dagher L, Furuse J, Geschwind JF, Ladron de Guevara L, Papandreou C, Sanyal AJ, Takayama T, Yoon SK, Nakajima K, Lehr R, Heldner S, Ye SL. Regional differences in sorafenib-treated patients with hepatocellular carcinoma: GIDEON observational study. Liver Int. 2016 Aug;36(8):1196-205. doi: 10.1111/liv.13096. Epub 2016 Apr 1. PMID 26901163
- [Derived] Lencioni R, Marrero J, Venook A, Ye SL, Kudo M. Design and rationale for the non-interventional Global Investigation of Therapeutic DEcisions in Hepatocellular Carcinoma and Of its Treatment with Sorafenib (GIDEON) study. Int J Clin Pract. 2010 Jul;64(8):1034-41. doi: 10.1111/j.1742-1241.2010.02414.x. PMID 20642705